CLINICAL TRIAL: NCT01012453
Title: Hand Eczema Trial: A Randomised Clinical Trial of the Effect of Classification and Individual Counselling Among Health Care Workers With Hand Eczema
Brief Title: A Randomised Clinical Trial in a Population of Health Care Workers With Hand Eczema
Acronym: HET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: The Danish Working Environment Authority (Unknown); Region Zealand (Other)
Responsible Party: Kristina Ibler MD, Ph.d student, Dermatological Department, Roskilde County Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SJ-126
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Eczema; Dermatitis; Skin Disease
Keywords: Hand eczema; Hand dermatitis; Occupational skin disease; skindisease in health care workers; occupational hand dermatitis; occupational hand eczema
MeSH Terms: conditions — Eczema; Dermatitis; Skin Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hand Eczema in health care workers (No Intervention)
  Interventions: Behavioral: A randomised clinical trial of the effect of classification and individual counselling

INTERVENTIONS:
Behavioral: A randomised clinical trial of the effect of classification and individual counselling — The trial to be conducted is a randomised single-blinded parallel study. It is divided in two stages, T = 0 and follow-up at T = 6 months. All included participants will have a clinical examination at the beginning and at follow-up in the trial. Half of the participants will be randomised to intervention, the other half to control. The participants in the intervention group will, after the first clinical examination, pass on directly to the intervention which includes an allergological examination (patch and prick testing). Three days later they will be examined by a physician who will interpret the patch test and give a thorough, individual guidance in skin protection and occupational safety. The clinical examination of all participants at follow-up will reveal the difference in outcomes in the intervention and the control group.

SUMMARY:
Objectives and perspective:

1. To estimate the prevalence of hand eczema in a cohort of health care workers and assess exposures in the hospital environment that can lead to hand eczema . To investigate the knowledge of skin protection among health care workers.
2. To classify subtypes of hand eczema, assess severity of hand eczema and quality of life in health care workers with hand eczema
3. To evaluate the effect of a combination of classification of hand eczema and individual work-related counseling in skin protective behavior.

The overall perspective of the trial is to develop new strategies for prevention of occupational hand eczema in health care workers.

Hypotheses:

* Irritant contact dermatitis is more common than allergic contact dermatitis.
* The combination of precise classification (subtyping of HE) and individual counseling will have a positive impact on the prognosis of hand eczema.
* The positive impact on the prognosis of hand eczema will have a positive impact on quality of life (QoL).
* The knowledge of protective behavior will increase.
* Education in a skin care program will have a positive impact on skin protective behavior.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited on the basis of the results from the questionnaire investigation of 3,181 HCW in three Danish hospitals in the same region. Participants who have answered "yes" to the validated question "Have you had hand eczema within the past twelve months?" will be invited to take part in the clinical trial.
* Informed written consent must be present in order to participate.

Exclusion Criteria:

* Pregnancy
* Systemic use of immunosuppressive drugs
* Systemic use of retinoids
* Active psoriatic lesions on the hands
* Any serious medical condition which, in the opinion of the investigator, may interfere with the evaluation of the results
* Lack of informed written consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Objective assessment of disease severity (HE), measured by HECSI-score at time = 6 months versus HECSI-score at time = 0. | 6 months

SECONDARY OUTCOMES:
Secondary outcomes: -Subjective assessment of disease severity (HE) -Number of eruptions through the past three months -Knowledge of skin protection -Skinprotective behaviour -Quality of life | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Holbaek Hospital, Holbæk
  - Koege Hospital, Koege
  - Dermatological Department, Roskilde County Hospital, Roskilde

REFERENCES:
- [Derived] Ibler KS, Jemec GB, Diepgen TL, Gluud C, Lindschou Hansen J, Winkel P, Thomsen SF, Agner T. Skin care education and individual counselling versus treatment as usual in healthcare workers with hand eczema: randomised clinical trial. BMJ. 2012 Dec 12;345:e7822. doi: 10.1136/bmj.e7822. PMID 23236031
- [Derived] Ibler KS, Agner T, Hansen JL, Gluud C. The Hand Eczema Trial (HET): Design of a randomised clinical trial of the effect of classification and individual counselling versus no intervention among health-care workers with hand eczema. BMC Dermatol. 2010 Aug 31;10:8. doi: 10.1186/1471-5945-10-8. PMID 20807407